CLINICAL TRIAL: NCT03784573
Title: Canine-Assisted Anxiety Reduction In Emergency Care
Acronym: CANINE III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Heather Kelker, Principal Investigator, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1811186507
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Anxiety; Opioid Use; Children; Therapy Dog
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized per dog and handler availability, but subjects that are excluded due to an aversion or dogs or per the Child Life staff member, can be in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dog + handler (Active Comparator)
  Interventions: Behavioral: Dog + handler
- No dog (Placebo Comparator)
  Interventions: Behavioral: No dog

INTERVENTIONS:
Behavioral: Dog + handler — Dog + handler
  Arms: Dog + handler
Behavioral: No dog — No dog
  Arms: No dog

SUMMARY:
Compare the effect of a single exposure to a therapy dog and handler within the pediatric emergency department patient with anxiety by measuring the change in patient perception of anxiety before and after dog exposure using the FACES scale. We will also measure galvanic skin response (resistance to electrical current).

DETAILED DESCRIPTION:
This study challenges current dogma by introducing a widely available, low cost method of dog therapy to reduce patient stress. The organization "Paws of Love" estimates that it has 180,000 volunteers who have qualified therapy dogs and who are generally willing to volunteer their time in emergency care. The benefits may include improved perception of wellness, less opioid use, and decreased use of physical and chemical restraints. As a further extrapolation, this secondary effect may extend to improved patient-doctor communication and patient experience. This will in turn improve patient safety in the Emergency Department, decreasing the number of adverse events, and decreasing the risk of medical malpractice by improving the patient-provider relationship. (6, 7)

ELIGIBILITY:
Inclusion Criteria:

* 4-17 years old;
* Physician or nurse with primary care responsibilities believes that the patients has a moderate to high level of anxiety

Exclusion Criteria:

- violent behavior and any reported prior fear or adverse reaction to dogs in the dog intervention group.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety level of subject | 45 minutes
  Change in anxiety level of subject with the use of the FACES scale

SECONDARY OUTCOMES:
Perception of anxiety level from physician | 60 minutes
  Change in perception anxiety level of subject with the use of the FACES scale
Perception of pain level from physician | 60 minutes
  Change in perception of pain level of subject with the use of a Wong-Baker Faces pain scale
Perception of anxiety level from parent(s) | 60 minutes
  Change in perception of anxiety level of subject by their parent(s) with the use of the FACES scale
Perception of pain level from parent(s) | 60 minutes
  Change in perception of pain level of subject by the parent(s) with the use of a Wong-Baker Faces pain scale
Meds | 4 hours
  Number of medications used to reduce anxiety in the different arms
Physical restrain use | 4 hours
  Number of times physical restraints are used

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Riley Children's Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Kelker HP, Siddiqui HK, Beck AM, Kline JA. Therapy Dogs for Anxiety in Children in the Emergency Department: A Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e250636. doi: 10.1001/jamanetworkopen.2025.0636. PMID 40085085